CLINICAL TRIAL: NCT05234827
Title: Effects Of Virtual Reality Based Rehabilitation Program On Physical Fitness In Patient With Chronic Obstructive Pulmonary Disorders
Brief Title: Virtual Reality Exercise on COPD Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC0872 Amna Syed
Record Dates: First submitted 2021-09-23; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: COPD
Keywords: physical fitness; Virtual reality; rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): VR sessions include a device (XBOX 360) and motion sensor (Kinect) and LED (tv screen) with speakers attached. Height of the device is 1m while tv screen is placed 2.5m away, motion sensor is placed 1.2m away from the patient, play area should be 1.8m wide and long. Instruction to play game is provided to each patient. Before starting each training session, the device was adjusted to correctly follow the movements of each patient. VR session includes games by Kinect Adventures (Microsoft games studios, Washington, US) which include minigames in which patients participated these mini games are 20000 Leaks, Curvy Creek, Rally Ball and Reflux Ridge.
  Interventions: Other: Virtual Reality; Other: Control
- Control (Active Comparator): Total time duration for session is 40 minutes in which 5 min of warm up exercises which include heel raises, arm circles, side leg raises, trunk rotation, elbow flexion and extension, knee flexion and extension, and shoulder internal and external rotation, 30 min of bicycling and after that 5-7 min of cool down exercises which include full body stretches i.e., toe touching, pectoralis major stretch, side by side bending, quadricep stretch, hamstring stretch, trapezius stretch and deep breathing
  Interventions: Other: Virtual Reality; Other: Control

INTERVENTIONS:
Other: Virtual Reality — Total time duration for session is 40 minutes which includes 5 min of warm exercises which include heel raises, arm circles, side leg raises, trunk rotation, elbow flexion and extension, knee flexion and extension, and shoulder internal and external rotation, 30 minutes of VR session and 5-7 min of cool down exercises which include full body stretches i.e., toe touching, pectoralis major stretch, side by side bending, quadricep stretch, hamstring stretch, trapezius stretch and deep breathing.
Other: Control — Control group receive endurance exercise testing in which stationary cycle is used for 30 min per session. It includes lower extremity strengthening i.e., increases hamstring and quadricep strength. Total time duration for session is 40 minutes in which 5 min of warm up exercises which include heel raises, arm circles, side leg raises, trunk rotation, elbow flexion and extension, knee flexion and extension, and shoulder internal and external rotation, 30 min of bicycling and after that 5-7 min of cool down exercises which include full body stretches i.e., toe touching, pectoralis major stretch, side by side bending, quadricep stretch, hamstring stretch, trapezius stretch and deep breathing.

SUMMARY:
The program allows the patient to interact with the simulated VR technology using motion sensors, focusing on patients' fitness through various tests providing them a clinically stable environment; to counter moderate level of diseases according to GOLD criteria and to monitor the effects of exercise program on dyspnea. The purpose of this study is to facilitate the patients so that they get acquainted with the digital technology with significant contribution towards pulmonary rehabilitation program for COPD patients. It also analysis the satisfaction of the patients and encourages the use of emerging technology integrated with clinical trials.

DETAILED DESCRIPTION:
Chronic obstructive lung disease (COPD) is a reversible lung disease which is a principal cause of morbidity and mortality worldwide. It is the third leading cause of death worldwide according to the reports of American Thoracic Society (ATS) and European- Respiratory Society. According to World Health Organization (WHO), every year death and in 2030 it will become the third most common cause of death. COPD risk factors includes smoking tobacco, exposure to dusts, hereditary predisposition, and fumes, indoor and outdoor air pollutants, ageing, and asthma. Out of all these risk factors, the main reason that develops COPD fastest is smoking which is further linked with depression

ELIGIBILITY:
Inclusion Criteria:

* Age:50-70 years
* Both genders
* Clinical Signs and Symptoms of Moderate COPD (GOLD Criteria)
* Clinically Stable
* Ratio of FEV1/ FVC is <0.7
* Reported Smoking History

Exclusion Criteria:

* Pneumonia, tuberculosis, and other respiratory
* inflammatory disease
* Heart Failure
* Advanced Uncontrolled Hypertension
* Post Cardiac or Thoracic Surgery (< 6 Months)
* Neuromuscular Disorders
* Metal Implant in Lower Limb
* Cardiac Pacemaker
* Cognitive Dysfunction or Mini-Mental Scale Scores <24
* Long- term Non-Invasive Ventilation
* Comorbidity that could Limit Exercise Testing and Training i.e., Arthritis, Osteoporosis, Fracture, Diabetic Neuropathy etc.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
30 Second Chair stand test (Senior Fitness Test Battery) | 0 week
  To measure the leg strength and endurance. The chair stand test is similar to a squat test to measure leg strength, in which participants stand up repeatedly from a chair for 30 seconds. Its category scoring based on the seconds, below average (<14), average (14 to 19) and above average (>19). Assessment done on baseline, 2nd week and fourth week.
30 Second Chair stand test (Senior Fitness Test Battery) | 2nd week
  To measure the leg strength and endurance. The chair stand test is similar to a squat test to measure leg strength, in which participants stand up repeatedly from a chair for 30 seconds. Its category scoring based on the seconds, below average (<14), average (14 to 19) and above average (>19).Assessment done on baseline, 2nd week and fourth week.
30 Second Chair stand test (Senior Fitness Test Battery) | 4th week
  To measure the leg strength and endurance. The chair stand test is similar to a squat test to measure leg strength, in which participants stand up repeatedly from a chair for 30 seconds. Its category scoring based on the seconds, below average (<14), average (14 to 19) and above average (>19).Assessment done on baseline, 2nd week and fourth week. Assessment done on baseline, 2nd week and 4th week.
Arm Curl Bicep Test(Senior Fitness Test Battery) | 0 week
  Test to measure the upper body strength and endurance. The aim of this test is to do as many arm curls as possible in 30 seconds. This test is conducted on the dominant arm side (or stronger side).5 pound weight (women, SFT), 8 pound weight (for men). A chair without armrests, stopwatch. The measurement according to complete in seconds below average (<16), average (16 to 22) and above average (>22). Assessment done on baseline, 2nd week and 4th week.
Arm Curl Bicep Test(Senior Fitness Test Battery) | 2nd week
  Test to measure the upper body strength and endurance. The aim of this test is to do as many arm curls as possible in 30 seconds. This test is conducted on the dominant arm side (or stronger side).5 pound weight (women, SFT), 8 pound weight (for men). A chair without armrests, stopwatch. The measurement according to complete in seconds below average (<16), average (16 to 22) and above average (>22). Assessment done on baseline, 2nd week and 4th week.
Arm Curl Bicep Test(Senior Fitness Test Battery) | 4th week
  Test to measure the upper body strength and endurance. The aim of this test is to do as many arm curls as possible in 30 seconds. This test is conducted on the dominant arm side (or stronger side).5 pound weight (women, SFT), 8 pound weight (for men). A chair without armrests, stopwatch. The measurement according to complete in seconds below average (<16), average (16 to 22) and above average (>22). Assessment done on baseline, 2nd week and 4th week.
Chair Sit & reach test(Senior Fitness Test Battery) | 0 week
  The Chair Sit and Reach test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors. This test measures lower body flexibility. The score is recorded to the nearest 1/2 inch or 1 cm as the distance reached, either a negative or positive score. Assessment done on baseline, 2nd week and 4th week.
Chair Sit & reach test(Senior Fitness Test Battery) | 2nd week
  The Chair Sit and Reach test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors. This test measures lower body flexibility. The score is recorded to the nearest 1/2 inch or 1 cm as the distance reached, either a negative or positive score. Assessment done on baseline, 2nd week and 4th week.
Chair Sit & reach test(Senior Fitness Test Battery) | 4th week
  The Chair Sit and Reach test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors. This test measures lower body flexibility. The score is recorded to the nearest 1/2 inch or 1 cm as the distance reached, either a negative or positive score. Assessment done on baseline, 2nd week and 4th week.
Back Scratch Test(Senior Fitness Test Battery) | 0 week
  The Scratch Test, measures how close the hands can be brought together behind the back. This test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors. This test measures general shoulder range of motion. Record the best score to the nearest centimeter or 1/2 inch. The higher the score the better the result. Below is a table showing the recommended ranges (in inches) for this test based on age groups (from Jones & Rikli, 2002). Assessment done on baseline, 2nd week and 4th week.
Back Scratch Test(Senior Fitness Test Battery) | 2nd week
  The Scratch Test, measures how close the hands can be brought together behind the back. This test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors. This test measures general shoulder range of motion. Record the best score to the nearest centimeter or 1/2 inch. The higher the score the better the result. Below is a table showing the recommended ranges (in inches) for this test based on age groups (from Jones & Rikli, 2002). Assessment done on baseline, 2nd week and 4th week.
Back Scratch Test(Senior Fitness Test Battery) | 4th week
  The Scratch Test, measures how close the hands can be brought together behind the back. This test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors. This test measures general shoulder range of motion. Record the best score to the nearest centimeter or 1/2 inch. The higher the score the better the result. Below is a table showing the recommended ranges (in inches) for this test based on age groups (from Jones & Rikli, 2002). Assessment done on baseline, 2nd week and 4th week.
8 Foot up & go test (Senior Fitness Test Battery) | 0 week
  The '8 Foot Up-and-Go' is a coordination and agility test for the elderly, which is part of the Senior Fitness Test Protocol. This test measures speed, agility and balance while moving. Take the best time of the two trails to the nearest 1/10th second. Below is a table showing the recommended ranges in seconds for this test based on age groups (from Jones & Rikli, 2002). Assessment done on baseline, 2nd week and 4th week.
8 Foot up & go test (Senior Fitness Test Battery) | 2nd week
  The '8 Foot Up-and-Go' is a coordination and agility test for the elderly, which is part of the Senior Fitness Test Protocol. This test measures speed, agility and balance while moving. Take the best time of the two trails to the nearest 1/10th second. Below is a table showing the recommended ranges in seconds for this test based on age groups (from Jones & Rikli, 2002). Assessment done on baseline, 2nd week and 4th week.
8 Foot up & go test (Senior Fitness Test Battery) | 4th week
  The '8 Foot Up-and-Go' is a coordination and agility test for the elderly, which is part of the Senior Fitness Test Protocol. This test measures speed, agility and balance while moving. Take the best time of the two trails to the nearest 1/10th second. Below is a table showing the recommended ranges in seconds for this test based on age groups (from Jones & Rikli, 2002). Assessment done on baseline, 2nd week and 4th week.
6 minute walk Test (Senior Fitness Test Battery) | 0 week
  The 6 Minute Walk test (6MWT) is designed to test the functional fitness of seniors. The aim of this test is to walk as quickly as possible for six minutes to cover as much ground as possible. measure the distance walked in 6 minutes to the nearest meter. The following regression equations were determined by Jenkins et al. (2009). Assessment done on baseline, 2nd week and 4th week.
  males: Walk Distance (meters) = 867 - (5.71 age, yrs) + (1.03 height, cm) females: Walk Distance (meters) = 525 - (2.86 age, yrs) + (2.71 height, cm) - (6.22 BMI)
6 minute walk Test (Senior Fitness Test Battery) | 2nd week
  The 6 Minute Walk test (6MWT) is designed to test the functional fitness of seniors. The aim of this test is to walk as quickly as possible for six minutes to cover as much ground as possible. measure the distance walked in 6 minutes to the nearest meter. The following regression equations were determined by Jenkins et al. (2009). Assessment done on baseline, 2nd week and 4th week.
  males: Walk Distance (meters) = 867 - (5.71 age, yrs) + (1.03 height, cm) females: Walk Distance (meters) = 525 - (2.86 age, yrs) + (2.71 height, cm) - (6.22 BMI)
6 minute walk Test (Senior Fitness Test Battery) | 4th week
  The 6 Minute Walk test (6MWT) is designed to test the functional fitness of seniors. The aim of this test is to walk as quickly as possible for six minutes to cover as much ground as possible. measure the distance walked in 6 minutes to the nearest meter. The following regression equations were determined by Jenkins et al. (2009). Assessment done on baseline, 2nd week and 4th week.
  males: Walk Distance (meters) = 867 - (5.71 age, yrs) + (1.03 height, cm) females: Walk Distance (meters) = 525 - (2.86 age, yrs) + (2.71 height, cm) - (6.22 BMI)
A Short Questionnaire for Satisfaction Evaluation of Virtual Rehabilitation Systems (USEQ) | 4th week
  It is necessary to evaluate the experience of individual whenever someone uses any system up to what extent user achieve goal with its effects and efficiency and satisfaction so that quality of user experience can be measure be and it is known as usability.(73) proper environment, product and instruction is required to obtain good usability of a system. One of the emerging technologies in the field of rehabilitation for different pathologies is virtual rehabilitation. Assessment done on 4th week.

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Al-Mustafa Trust Medical Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutkowski S, Rutkowska A, Kiper P, Jastrzebski D, Racheniuk H, Turolla A, Szczegielniak J, Casaburi R. Virtual Reality Rehabilitation in Patients with Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Jan 13;15:117-124. doi: 10.2147/COPD.S223592. eCollection 2020. PMID 32021150
- [Background] Nafees AA, Fatmi Z, Kadir MM, Sathiakumar N. Chronic Bronchitis and Chronic Obstructive Pulmonary Disease (COPD) Among Textile Workers in Karachi, Pakistan. J Coll Physicians Surg Pak. 2016 May;26(5):384-9. PMID 27225143
- [Background] Rutkowski S, Szczegielniak J, Szczepanska-Gieracha J. Evaluation of the Efficacy of Immersive Virtual Reality Therapy as a Method Supporting Pulmonary Rehabilitation: A Randomized Controlled Trial. J Clin Med. 2021 Jan 18;10(2):352. doi: 10.3390/jcm10020352. PMID 33477733